CLINICAL TRIAL: NCT04465695
Title: An Open-label Randomised Controlled Trial on Dual Therapy With Interferon Beta-1b and Clofazimine Combination, as Treatment for COVID-19 Infection
Brief Title: Dual Therapy With Interferon Beta-1b and Clofazimine for COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ivan FN Hung MD, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-463
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: COVID-19; hospitalised; IFN beta-1b; clofazimine
MeSH Terms: conditions — COVID-19 | interventions — Interferon beta-1b; Clofazimine

STUDY DESIGN:
Intervention Model Description: Open-label randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IFN beta-1b and clofazimine (Experimental): A 3-day course of 3 doses of subcutaneous injection of interferon β-1b 1mL (0.5mg; 16 million IU) consecutively on day 1 to day 3 and oral clofazimine 100mg twice daily on day 1, then 100mg daily for 2 days plus standard care
  Interventions: Drug: Interferon beta-1b; Drug: Clofazimine
- Clofazimine (Active Comparator): A 3-day course of oral clofazimine 100mg twice daily on day 1, then 100mg daily for 2 days plus standard care
  Interventions: Drug: Clofazimine
- Control (No Intervention): Standard care alone

INTERVENTIONS:
Drug: Interferon beta-1b — Subcutaneous injection of interferon β-1b 1mL (0.5mg; 16 million IU) for 3 days
  Arms: IFN beta-1b and clofazimine
Drug: Clofazimine — Oral 100mg twice daily on day 1, then 100mg daily for 2 days
  Arms: Clofazimine; IFN beta-1b and clofazimine

SUMMARY:
To conduct an open-label randomized controlled trial on a short course of interferon β-1b and clofazimine combination treatment for patients hospitalized for COVID-19 infection. To assess its safety and clinical efficacy.

DETAILED DESCRIPTION:
The novel coronavirus (SARS-CoV-2), is a single-stranded RNA coronavirus. The virus was first isolated from patients presented with pneumonia in Wuhan in December 2019.Sequences of the Wuhan betacoronavirus show similarities to betacoronaviruses found in bats, sharing a common ancestor with the 2003 SARS coronavirus (SARS-CoV) and the bat coronavirus HKU9-1, a virus found in fruit bats. Similar to SARS-CoV, it is a member of Beta-CoV lineage B. Five genomes of the novel coronavirus have been initially isolated and reported including BetaCoV/Wuhan/IVDC-HB-01/2019, BetaCoV/Wuhan/IVDC-HB-04/2020, BetaCoV/Wuhan/IVDC-HB-05/2019, BetaCoV/Wuhan/WIV04/2019, and BetaCoV/Wuhan/IPBCAMS-WH-01/2019 from the China CDC.

The SARS-CoV-2 has since spread from China to the rest of the world. As of 1 July 2020, more than 10 million people been confirmed to have infected by SARS-CoV-2, resulting in more than 500,000 deaths. No specific antiviral treatment for the SARS-CoV-2 is currently available, but existing medication could be repurposed.

Genetic sequencing demonstrated similarity of the SARS-CoV-2 to the SARS-CoV and MERS CoV.2 We expect patients infected with the SARS-CoV-2 will also present similarly with initial upper respiratory tract symptoms including fever, cough, sputum, myalgia and shortness or breath. More severe cases might complicate with pneumonia and required ventilatory or ECMO support. According to our previous studies in 2003 on patients hospitalized for severe SARS-CoV, the viral load peaked between day 7 from symptoms onset and coincided with clinical deterioration of pneumonia and respiratory failure, with majority of the patients required intensive care support. Higher viral load isolated from different human system also correlated with worsened SARS manifestation and complications.

Previously, the investigators have demonstrated that interferon β-1b, commonly used in the treatment of multiple sclerosis and lopinavir/ ritonavir, also demonstrated to improve the outcome of MERS-CoV infection in a non-human primate model of common marmoset.7

More recently, the investigators have demonstrated that the triple combination of interferon β-1b, lopinavir/ ritonavir and ribavirin was significantly more effective in alleviating symptoms and respiratory SARS-CoV-2 viral load than lopinavir/ ritonavir with ribavirin or lopinavir/ ritonavir alone, suggesting that interferon β-1b might be the most potent antiviral among the three.

Another in-vitro study on an oral antimicrobial clofazimine for treatment of non-tuberculous mycobacterium infection has been proven to reduce SARS-CoV-2 viral load.

Therefore, the investigators propose to perform a prospective open-label randomised controlled trial among adult patients hospitalised after July 2020 for virologically confirmed SARS-CoV-2 infection. Patients will be randomly assigned to one of the three groups: group A: a 3-day course of 3 doses of subcutaneous injection of interferon β-1b 1mL (0.5mg; 16 million IU) consecutively on day 1 to day 3 and oral clofazimine 100mg twice daily on day 1, then 100mg daily for 2 days plus standard care, or group B: oral clofazimine 100mg twice daily on day 1, then 100mg daily for 2 days plus standard care, or group C: standard care alone (1:1:1).

ELIGIBILITY:
Inclusion Criteria:

1. Recruited subjects include all adult patients 18 years or above hospitalized for virologic confirmed SARS-CoV-2 infection.
2. All subjects give written informed consent. For patients who are critically ill, requiring ICU, ventilation or confused, informed consent will be obtained from spouse, next-of-kin or legal guardians.
3. Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures.
2. Allergy or severe reactions to the study drugs
3. Patients taking medication that will potentially interact with l interferon beta-1b or clofazimine
4. Patients with known history of severe depression
5. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to recruitment in this study or expect to receive an experimental agent during this study.
6. To participate in an unrelated trial during the current clinical trial. Nevertheless, the patients have the right to withdraw from the current clinical trial to join another clinical trial.
7. Have a history of alcohol or drug abuse in the last 5 years.
8. Have any condition that the investigator believes may interfere with successful completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical alleviation of symptoms | 7 days
  Time to complete alleviation of symptoms as defined by NEWS of 0 maintained for 24 hours

SECONDARY OUTCOMES:
Hospitalisation | 14 days
  Length of hospitalisation
Time to negative viral load | 7 days
  Time to negative nasopharyngeal swab, throat saliva and sputum viral load by RT-PCR
Inflammatory changes | 7 days
  Cytokine/ chemokine changes
Mortality | 30 days
  One month mortality rate
Adverse events | 30 days
  Adverse events during and shortly after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — HKU
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
To share anonymised participant data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 12 months of study published
Access Criteria: To be approved by the HKU/ IRB clinical trial study panel of valid research purpose

REFERENCES:
- [Background] Hung IF, Lung KC, Tso EY, Liu R, Chung TW, Chu MY, Ng YY, Lo J, Chan J, Tam AR, Shum HP, Chan V, Wu AK, Sin KM, Leung WS, Law WL, Lung DC, Sin S, Yeung P, Yip CC, Zhang RR, Fung AY, Yan EY, Leung KH, Ip JD, Chu AW, Chan WM, Ng AC, Lee R, Fung K, Yeung A, Wu TC, Chan JW, Yan WW, Chan WM, Chan JF, Lie AK, Tsang OT, Cheng VC, Que TL, Lau CS, Chan KH, To KK, Yuen KY. Triple combination of interferon beta-1b, lopinavir-ritonavir, and ribavirin in the treatment of patients admitted to hospital with COVID-19: an open-label, randomised, phase 2 trial. Lancet. 2020 May 30;395(10238):1695-1704. doi: 10.1016/S0140-6736(20)31042-4. Epub 2020 May 10. PMID 32401715
- [Background] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Background] Chu H, Chan JF, Wang Y, Yuen TT, Chai Y, Hou Y, Shuai H, Yang D, Hu B, Huang X, Zhang X, Cai JP, Zhou J, Yuan S, Kok KH, To KK, Chan IH, Zhang AJ, Sit KY, Au WK, Yuen KY. Comparative Replication and Immune Activation Profiles of SARS-CoV-2 and SARS-CoV in Human Lungs: An Ex Vivo Study With Implications for the Pathogenesis of COVID-19. Clin Infect Dis. 2020 Sep 12;71(6):1400-1409. doi: 10.1093/cid/ciaa410. PMID 32270184
- [Background] Chan JF, Yao Y, Yeung ML, Deng W, Bao L, Jia L, Li F, Xiao C, Gao H, Yu P, Cai JP, Chu H, Zhou J, Chen H, Qin C, Yuen KY. Treatment With Lopinavir/Ritonavir or Interferon-beta1b Improves Outcome of MERS-CoV Infection in a Nonhuman Primate Model of Common Marmoset. J Infect Dis. 2015 Dec 15;212(12):1904-13. doi: 10.1093/infdis/jiv392. Epub 2015 Jul 21. PMID 26198719
- [Background] Yuan S, Chan CC, Chik KK, Tsang JO, Liang R, Cao J, Tang K, Cai JP, Ye ZW, Yin F, To KK, Chu H, Jin DY, Hung IF, Yuen KY, Chan JF. Broad-Spectrum Host-Based Antivirals Targeting the Interferon and Lipogenesis Pathways as Potential Treatment Options for the Pandemic Coronavirus Disease 2019 (COVID-19). Viruses. 2020 Jun 10;12(6):628. doi: 10.3390/v12060628. PMID 32532085